CLINICAL TRIAL: NCT04892589
Title: The Role of the Proprioceptive Training in Functional Recovery of Patient With Thumb Base Osteoarthritis. A Multicenter Experimental Study
Brief Title: The Role of the Proprioceptive Training in Functional Recovery of Patient With Thumb Base Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Universitaria Reina Fabiola, Universidad Catolica de Cordoba (Other)
Responsible Party: Principal Investigator, Alejandra Tuljak, principal investigator, Clinica Universitaria Reina Fabiola, Universidad Catolica de Cordoba
Other Study IDs: 2021
Record Dates: First submitted 2021-04-30; First posted 2021-05-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Thumb Osteoarthritis
Keywords: Thumb pain; Thumb proprioception; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active Comparator: Control group: Thumb orthosis at night and day for 3 to 4 hours during Activities of Daily Living that included thumb metacarpophalangeal joint (MCP) for three months. In addition to a classic home exercise program.
- Experimental: Experimental group: The experimental group will receive thumb orthosis at night and daytime use for 3 to 4 hours during Activities of Daily Living that included the thumb MCP for three months. In addition to a classic home exercise program and a proprioceptive home exercises program divided in three phases.
  Interventions: Other: Proprioceptive thumb exercises.

INTERVENTIONS:
Other: Proprioceptive thumb exercises. — Exercises for recognition of thumb position and thumb force sense.
  Groups: Experimental: Experimental group

SUMMARY:
Diseases that have implications for the thumb impact its function, and consequently, people occupational performance. Carpometacarpal joint (CMC) thumb degeneration translates into osteoarthritis (OA). Joint congruence, ligament integrity and compression of the joint surfaces caused by muscle contraction have historically been considered the three basic pillars for carpus stability. In recent years, a new factor has been proposed to explain carpal stabilization mechanisms: proprioception. The dorsal ligament complex is the structure with the highest concentration of mechanoreceptors, especially Ruffini's corpuscles. This study aims to detect the effect of proprioceptive training on the functional recovery of people with CMC osteoarthritis in conservative treatments.

DETAILED DESCRIPTION:
The carpometacarpal joint (CMC) of the thumb presents a paradoxical relationship between mobility and stability that confers it a high mechanical complexity, and it is continuously subjected to great efforts and repetitive movements during its use that lead to degenerative changes in susceptible individuals. The thumb CMC join degeneration results in osteoarthritis (OA).

Joint congruence, ligament integrity, and compression of the articular surfaces caused by muscle contraction have historically been considered the three basic pillars for carpal stability. In recent years, a new factor has been proposed to explain carpal stabilization mechanisms: proprioception. All afferents originating from the thumb mechanoreceptors constitute thumb proprioception. The dorsal ligament complex is the structure with the highest concentration of mechanoreceptors, especially Ruffini's corpuscles.

Classically, in conservative treatments, orthotic positioning is paramount. This study aims to detect the effect of proprioceptive training on the functional recovery of people with CMC osteoarthritis, from the comparison of a classic conservative orthotic treatment protocol vs. a conservative orthotic treatment protocol including exercises for proprioceptive training.

A randomized clinical trial is proposed within a multicenter study involving the Clínica Universitaria Reina Fabiola, Argentina and the Centro Tecan. Clínica de la Mano, Spain. The patients will be randomized into a control group that will receive orthosis treatment; and an experimental group that will also receive a home proprioceptive exercise program. Pain will be evaluated with the Visual Analogue Scale; functional capacity with the Australian Canadian Osteoarthritis Hand Index Version Functional Subscale; Occupational Productivity Performance with the Canadian Measure of Occupational Performance; and proprioception with the Joint Position Sense Test. Follow up: at 30 days and at 90 days. 50 patients will participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade I, II or III thumb CMC joint OA in their dominant hand according to the Eaton Classification Stage
* Pain rating of 4/10 on the Visual Analogue Scale (VAS) during activities of daily living (ADLs) at the time of the therapy initial evaluation.
* The ability to read and understand the patient information sheets and exercises.
* A minimum thumb abduction capacity of 40º.

Exclusion Criteria:

* Previous hand and wrist surgeries, neurological disorders, diagnosis of OA that includes the wrist, rheumatoid arthritis, or any implication of an osteomyoarticular nature in the hand and / or wrist other than the CMC OA.
* Had received specific treatment for hand or thumb pain in the same limb in the last 6 months including an intra-articular joint injection to wrist, fingers, or thumb.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with carpometacarpal osteoarthritis of the thumb who require conservative treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline pain at 4 weeks.
  Visual Analogue Scale has been shown to be a reliable and valid instrument for pain assessment which is used frequently for clinical and research purposes. It consists of a 10-cm line anchored at each end. The left-hand anchor reads 'no pain' score 0 and the right-hand anchor reads 'worst possible pain' score 10; the patients marked a line to represent their pain level.
Visual Analogue Scale (VAS) | Change from 4 weeks pain at 12 weeks.
  Visual Analogue Scale has been shown to be a reliable and valid instrument for pain assessment which is used frequently for clinical and research purposes. It consists of a 10-cm line anchored at each end. The left-hand anchor reads 'no pain' score 0 and the right-hand anchor reads 'worst possible pain' score 10; the patients marked a line to represent their pain level.
Australian Canadian Osteoarthritis Hand Index version (AUSCAN) | Change from baseline hand function at 4 weeks.
  To assess the affection of the hands in rheumatic diseases, with good discriminatory capacity The functional capacity assessment subscale will be used, which provides specific data on the subject's ability to open / close water taps; turn the door handles / knobs; buttoning up; fastening / unbuttoning jewelry; open a new bottle; load a full pot; peel fruits and vegetables; lift large and heavy objects; wring out wet clothes / sponges or rags. This functional subscale evaluates from 9 to 45, with 9 being "no difficulty" and 45 "extreme difficulty"
Australian Canadian Osteoarthritis Hand Index version (AUSCAN) | Change from 4 weeks hand function at 12 weeks.
  To assess the affection of the hands in rheumatic diseases, with good discriminatory capacity The functional capacity assessment subscale will be used, which provides specific data on the subject's ability to open / close water taps; turn the door handles / knobs; buttoning up; fastening / unbuttoning jewelry; open a new bottle; load a full pot; peel fruits and vegetables; lift large and heavy objects; wring out wet clothes / sponges or rags. This functional subscale evaluates from 9 to 45, with 9 being "no difficulty" and 45 "extreme difficulty"

SECONDARY OUTCOMES:
Joint position Sense (JPS) | baseline-4 and 12 weeks
  Proprioception using active joint position sense (JPS) has been utilized in studies to establish a correlation between therapy intervention and proprioception. The target position of 30 degree CMC abduction will be selected. Joint angle will be measured using a standard clear plastic goniometer.
Canadian Occupational Performance Measure | baseline-4 and 12 weeks
  Patient's occupational performance will be measured with the Canadian Occupational Performance Measure (COPM).
  The COPM enables subjects to identify goals for hand therapy and engage in a subject-specific therapeutic process. It has been established that the COPM has good convergent validity and responsiveness for evaluating the relationship between patient self-perception and satisfaction for patients with CMC thumb OA .
Force Sense | baseline-4 and 12 weeks
  Patient's sensation force will be measured with the Force Sense.

CONTACTS AND LOCATIONS:
Locations (2):
- Clínica Universitaria Reina Fabiola, Córdoba, Argentina
- Centro TECAN Clinica de la Mano, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No